CLINICAL TRIAL: NCT02192528
Title: 25-Hydroxyvitamin D, 1,25-Dihydroxyvitamin D and Postoperative Outcome in Cardiac Surgical Patients
Brief Title: Vitamin D and Outcome in Cardiac Surgery
Acronym: Calcitop
Status: Completed | Type: Observational
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Sponsor
Other Study IDs: 008
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2014-07

CONDITIONS: Cardiovascular Disease
Keywords: vitamin D; 25-hydroxyvitamin D; 1,25-dihydroxyvitamin D; MACCE; mortality; cardiac; cerebrovascular
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cardiac surgical patients: patients undergoing a cardiac surgical procedure

SUMMARY:
We will use a retrospective data analysis to evaluate the association of the two vitamin D metabolites 25-hydroxyvitamin D and 1,25-dihydroxyvitamin D with clinical outcome in cardiac surgical patients. The occurrence of several postoperative adverse events such as myocardial infarction, low cardiac output syndrome, stroke and in-hospital death will be assessed from cardiac surgery to discharge. In addition, we will assess the association of the two vitamin D metaboolites with the duration of mechanical ventilatory support and intensive care unit stay from cardiac surgery to discharge. Moreover, in-hospital stay will be assessed according to vitamin D metabolite levels.

DETAILED DESCRIPTION:
In a retrospective data analysis, we will evaluate the association of vitamin D metabolites (circulating 25-hydroxyvitamin D and 1,25-dihydroxyvitamin D) with MACCE (major cardiac or cerebrovascular event) in cardiac surgical patients. The occurrence of several postoperative adverse events such as myocardial infarction, low cardiac output syndrome, stroke and in-hospital death will be assessed from cardiac surgery to discharge. Approximately 4,000 data sets from mid of 2012 until the end of 2013 will be analyzed. In all patients, we will also assess the association of vitamin D metabolite levels with the duration of mechanical ventilatory support and intensive care unit stay from cardiac surgery to discharge. Moreover, in-hospital stay will be assessed according to vitamin D status

ELIGIBILITY:
Inclusion Criteria:

* cardiac surgical patients aged 18 years and older

Exclusion Criteria:

* age < 18 years
* heart transplant recipients
* pacemaker or defibrillator implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cardiac surgical patients
Sampling Method: Probability Sample
Enrollment: 3852 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
major cardiac or cerebrovascular event (MACCE) | Patients will be followed for an average time of 14 days from cardiac surgery to discharge
  MACCE is defined as in-hospital death, myocardial infarction, low cardiac output syndrome or stroke.

SECONDARY OUTCOMES:
duration of ventilatory support | Patients will be followed for an average time of 14 days from cardiac surgery to discharge
intensive care unit stay | Patients will be followed for an average time of 14 days from cardiac surgery to discharge
in-hospital stay | Patients will be followed for an average time of 14 days from cardiac surgery to discharge
infection | Patients will be followed for an average time of 14 days from cardiac surgery to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Armin Zittermann, PhD, Principal Investigator — Heart & Diabetes Center North-Rhine Westfalia, Germany
Locations (1):
- Heart & Diabetes Center North-Rhine Westphalia, Bad Oeynhausen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zittermann A, Kuhn J, Dreier J, Knabbe C, Gummert JF, Borgermann J. Vitamin D status and the risk of major adverse cardiac and cerebrovascular events in cardiac surgery. Eur Heart J. 2013 May;34(18):1358-64. doi: 10.1093/eurheartj/ehs468. Epub 2013 Jan 12. PMID 23315905